CLINICAL TRIAL: NCT07046949
Title: A Randomized Controlled Double-blinded Trial Evaluating the Efficacy of the Anterior Quadratus Lumborum Block as a Component of Multimodal Perioperative Analgesia for Abdominal Hysterectomies
Brief Title: Anterior Quadratus Lumborum Block as a Component of Multimodal Analgesia for Abdominal Hysterectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuri Semenyuk Rivne Regional Clinical Hospital (Other)
Collaborators: Danylo Halytsky Lviv National Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7-A/2812
Record Dates: First submitted 2025-05-29; First posted 2025-07-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Uterine Bleeding; Uterine Neoplasms; Uterine Diseases; Uterine Fibroids
Keywords: Regional anesthesia; Quadratus lumborum block; Abdominal hysterectomy; Pain scores; Multimodal analgesia; Acute pain; Chronic pain; Pain management; Opioid consumption; Quality of recovery; Postoperative nausea and vomiting; General anesthesia; Blended anesthesia; Hemodynamics after surgery
MeSH Terms: conditions — Uterine Hemorrhage; Uterine Neoplasms; Uterine Diseases; Leiomyoma; Acute Pain; Chronic Pain; Agnosia; Postoperative Nausea and Vomiting | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: A two-arm parallel group design in which participants are randomly allocated to receive either general anesthesia and multimodal analgesia without QL-block or general anesthesia and multimodal analgesia including QL-block.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (control) (Active Comparator): Patients in Group I will undergo general anesthesia with tracheal intubation and mechanical ventilation. Analgesia regimen will include parenteral medication.
  Interventions: Drug: Parenteral administration of analgesics; Procedure: General Anesthesia (GA)
- Group II (QL) (Experimental): Patients in Group II (QL) will undergo general anesthesia with tracheal intubation and mechanical ventilation. Analgesia regimen will include parenteral medication and anterior quadratus lumborum block as a regional component.
  Interventions: Procedure: ANTERİOR QUADRATUS LUMBORUM BLOCK; Drug: Parenteral administration of analgesics; Procedure: General Anesthesia (GA)

INTERVENTIONS:
Procedure: ANTERİOR QUADRATUS LUMBORUM BLOCK — Ultrasound-guided anterior QL block performed preoperatively
  Arms: Group II (QL)
Drug: Parenteral administration of analgesics — Intravenous opioids or NSAIDs used perioperatively.
Procedure: General Anesthesia (GA) — Standard general anesthesia per continious 1% propofol infusion and propofol bolus administration, atracurium and fentanyl administration.

SUMMARY:
The main goal of this randomised double-blinded controlled trial is to assess whether adding anterior quadratus lumborum block preoperatively can reduce intraoperative and postoperative opioid consumption, reduce pain after abdominal hysterectomy and improve quality of recovery after anesthesia. The study hypothesis is that anterior QL block bilaterally before the start of a surgery has no impact on perioperative pain relief, can't reduce the need in opioids and will not improve quality of recovery after anesthesia.

All patients will undergo general anesthesia with tracheal intubation and mechanical ventilation. Patients will be randomized into two groups. In addition to general anesthesia and multimodal analgesia with parenteral medication II (QL) group will receive also anterior quadratus lumborum block as a regional component.

DETAILED DESCRIPTION:
Primary outcomes : intraoperative fentanyl consumption, daily requirement of morphine and pain level (with visual analogue scale - VAS) after surgery. Secondary outcomes: quality of recovery after anesthesia (with QoR-15 questionnaire), heart rate perioperatively, mean arterial pressure perioperatively, incidence of postoperative nausea.

Thromboprophylaxis will be administered based on the risk of thromboembolic complications for all patients. In the operative room all patients will receive ondansetron, dexamethasone and tranexamic acid. Patients will be told that they will receive multimodal analgesia but they won't know if they get a regional component (quadratus lumborum block). The randomisation will take place in the operative room. After general anesthesia induction and endotracheal intubation attending anesthesiologist will leave the operative room and anesthesiologist-resident will perform randomization and QL-block or won't perform QL-block. Thus participants and attending anesthesiologist won't know the randomisation result. In our study attending anaesthesiologist will be the researcher who will collect and analyse data. After the intubation patients of the control group will receive acetaminophen 1000 mg, dexketoprofen 50 mg before incision and MgSO4 1250 mg with ongoing continuous infusion of MgSO4 2500 mg per hour. In addition to these analgesia regimen patients in the II (QL) group will receive bilateral ultrasound-navigated anterior quadratus lumborum block before the start of the surgery. The investigators will use a convex low-frequency transducer with a frequency of 1.5-5 Mhz (General Electric Logiq e ultrasound machine). The block will be performed in the patient's spine position. Investigators choose anterior approach hypothesizing its superiority over other approaches to quadratus lumborum block. After proper visualization and obtaining an adequate sonographic image, the 22g needle will be inserted through the lateral abdominal wall and will be advanced through the skin, subcutaneous fat tissue, external oblique muscle, internal oblique muscle, aponeurosis of the transverse abdominis muscle, then it will be advanced through the quadratus lumborum muscle and operator will reach thoracolumbar fascia, between the quadratus lumborum muscle and the psoas major muscle. In this localization anesthesiologist-resident will inject a local anesthetic. Operator will use 20 ml of 0,25% bupivacaine with 4 mg of dexamethasone as adjuvant for one side, all blocks will be performed bilaterally only. General anaesthesia will be maintained by continuous propofol infusion with target effect site concentration 3-3,5 mcg/ml, atracurium infusion with target effect site concentration 900 ng/ml and bolus fentanyl injections to maintain target effect site concentration 2-4 ng/ml. All target concentrations will be calculated via ITIVA version 6.3.2 software. Attending anesthesiologist will modify the dosage of anesthetic drugs, particularly fentanyl, reducing them if necessary. At postoperative stage for patients of both groups investigators plan to administer multimodal analgesia: dexketoprofen (150 mg/day), acetaminophene (4000 mg/day). In addition, in the case of severe pain - morphine will be added (5-20 mg/day).

Mechanical ventilation will be performed in pressure-regulated volume control ventilation mode counting tidal volume 6 ml/kg (Getinge Flow-e anesthesia machine). Intraoperatively attending anesthesiologist will count the fentanyl consumption considering that the length of the surgeries will not have significant differences.

At the end of the surgery investigators will count total amount of administered fentanyl, evaluate heart rate and mean arterial pressure.

After the end of the surgeries patients will be extubated and transferred to the postoperative ward. After the surgery investigators are planning to evaluate morphine consumption, level of pain according to the visual analogue scale (VAS), quality of recovery after anesthesia (with QoR-15 questionnaire), heart rate, mean arterial pressure, incidences of nausea.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA status I-II
* patients with symptomatic fibroids
* patients scheduled for abdominl hysterectomy

Exclusion Criteria:

* refusal to participate in the study at any of its stages
* ASA class ≥ III
* body mass index > 40 kg/m2
* use of opiate receptor agonists/antagonists before surgery
* uncontrolled hypertension

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Pain level after surgery | It will be checked at the folowing stages of the study: 30 minutes (m30) 6 hours (h6), 12 hours (h12), 24 hours (h24), 48 hours (h48) after the end of the surgery.
  It will be tested using visual analogue scale (VAS)
Requirement of morphine for 24 hours | 24 hours (h24), 48 hours (h48) after the surgery
  The investigators will count a dose of morphine administered for patients of both groups postoperatively
Intraoperative fentanyl consumption | Intraoperative stage, at the end of the surgery (h0)
  The investigators will compare fentanyl consumption between two groups, considering that the duration of surgeries differences won't be statistically significant.

SECONDARY OUTCOMES:
Quality of recovery after anesthesia | The investigators will test it in 24 hours after the end of the surgery (h24)
  The investigators will measure it using QoR-15 questionnaire
Postoperative nausea | At 30 minutes (m30), 6 hours (h6), 12 hours (h12), 24 hours (h24) after the end of the surgery
  The investigators will define the incidents of nausea in both groups after the surgery
Perioperative heart rate | The investigators will evaluate parameters at intraoperative stage (h0), 30 minutes (m30), 6 hours (h6), 12 hours (h12), 24 hours (h24), 48 hours (h48) after the surgery.
  The investigators will evaluate heart rate during the surgery and after it will be finished.
Mean arterial pressure perioperatively | The investigators will evaluate the parameters at intraoperative stage (h0), 30 minutes (m30), 6 hours (h6), 12 hours (h12), 24 hours (h24), 48 hours (h48) after the surgery.
  The investigators will evaluate mean arterial pressure during the surgery and after it will be finished.

CONTACTS AND LOCATIONS:
Overall Officials: Olha Filyk, Professor, Study Chair — Danylo Halytsky Lviv National Medical University
Locations (1):
- Yuri Semenyuk Rivne regional cinical hospital, Rivne, Rivne Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared.